CLINICAL TRIAL: NCT07116421
Title: Effect of 2-phenylethanol Odor Exposure on Ictal Apneic Episode Occurrence Rate in Patients With Epilepsy
Brief Title: Effect of Rose Odor Exposure on Ictal Apnea
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, William P. Nobis, Assistant Professor of Neurology, Vanderbilt University Medical Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 241251
Record Dates: First submitted 2025-08-06; First posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Epilepsy; Sudden Unexpected Death in Epilepsy
Keywords: SUDEP; Epilepsy; Sudden Unexpected Death in Epilepsy
MeSH Terms: conditions — Epilepsy; Sudden Unexpected Death in Epilepsy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rose scent exposure (Experimental): Ambient rose scent exposure via aromatherapy diffuser into patient room for 24 hours
  Interventions: Drug: 2-phenylethanol rose scent
- Room air (No Intervention): Scentless room air for 24 hours

INTERVENTIONS:
Drug: 2-phenylethanol rose scent — Name: 2-phenylethanol (rose scent). Dose: 3 drops, diffused into room air over 24 hours. Frequency: Once over 24 hours. Route of administration: Essential oil diffuser. Manufactured by: The Essential Oil Company in Portland, OR. Manufacturing details: The rose scent is purified by hydrodistillation, shelf-stable, and in terms of verification of quality has been previously used in a peer-reviewed and IRB-approved study by Woo et al (2023) published in Frontiers in Neuroscience. Preparation: The Key Personnel listed in the study's IRB will prepare the rose essential oil scent by squeezing 3 drops of the product from the manufactured bottle into the essential oil compartment of the "Aroma Ace™ MINI Diffuser" essential oil diffuser, corresponding with both the rose essential oil and diffuser manufacturers' instructions for each product respectively.
  Other Names: Rose aromatherapy; Rose smell; Rose oil; Rose diffusor scent
  Arms: Rose scent exposure

SUMMARY:
This study will investigate the potential benefits of rose scent in reducing the risk of Sudden Unexpected Death in Epilepsy (SUDEP) in patients with epilepsy. Participants will engage in their routine inpatient observational EEG monitoring for 24 hours followed by an additional 24 hours of observational EEG monitoring with continuous exposure to rose scent, during which an essential oil diffusor with rose scent will be placed in their hospital room. During these 48 total hours of the study, participants will wear a respiratory monitoring belt across their upper chest to measure their breathing.

Potential risks include distress or discomfort when smelling the rose scent used in the study, a physical reaction to the rose scent, and discomfort or feelings of restrictiveness when wearing the respiratory monitoring belt. The total time commitment of the study is 48 consecutive hours over the course of the participants' inpatient EMU stay, during which there will be no restrictions on daily activities during the standard inpatient EMU admission except that participants must wear their respiratory belt for a majority of this 2-day period.

DETAILED DESCRIPTION:
[1.0. Background] Sudden unexpected death in epilepsy (SUDEP) affects 1 in 1000 patients with epilepsy every year.1 SUDEP is thought to occur due to respiratory dysfunction during seizure periods, but the exact mechanism remains unclear. Medical management to treat and prevent SUDEP is thus limited and warrants further investigation.

[2.0. Rationale and Specific Aims] Our aim is to observe seizure activity and respiratory function via EEG and respiratory monitoring belt, respectively, following 24 hours of exposure to rose scent via essential oil diffusor in adult patients with epilepsy who have been admitted to the epilepsy monitoring unit (EMU) for observation without medication changes. We hope to uncover a potential olfactory intervention for SUDEP in adult epilepsy patients that would build a stronger understanding of the pathophysiology behind the condition and help reduce the risk of death due to SUDEP.

[3.0. Animal Studies and Previous Human Studies] Several human studies have uncovered a general connection between olfactory modulation and epilepsy by exposing participants with epilepsy to certain scents and then measuring either the frequency and duration of their seizure activity or their EEG activity following scent exposure. A prior human study conducted by Yilmaz et al. indicated a significant antiepileptic benefit of olfactory modulation using lavender scent in 28 pediatric and adult patients aged 8-65 years with drug-resistant epilepsy.6 Focusing on the relationship between olfactory modulation and SUDEP specifically, the principle investigator of this study, Dr. Nobis, has conducted preliminary animal studies indicating that Dravet Syndrome mouse models, which exhibit spontaneous seizures and high SUDEP rates due to a heterozygous deletion in the scn1a gene (scn1a +/-), demonstrate reduced mortality when exposed to 2-phenylethanol (2PE, the major component of rose scent).

[4.0. Inclusion/Exclusion Criteria]

Inclusion Criteria.

* Adult epilepsy patients over the age of 18
* Admission to the inpatient epilepsy monitoring unit (EMU) at Vanderbilt University Medical Center (VUMC)
* Undergoing observational EEG monitoring without treatment involving seizure medication changes or other interventions for at least 48 hours Exclusion Criteria.
* Patients under the age of 18
* Patients receiving EEG monitoring without interventions from baseline for less than 48 hours
* Patients who are not receiving EEG monitoring as a part of their inpatient admission.

[5.0. Enrollment/Randomization] Resident fellow physician staff in the Epilepsy Division of the Department of Neurology at Vanderbilt University Medical Center will identify prospective participants on a rolling basis in the inpatient epilepsy monitoring unit. Key study personnel will then visit prospective participants in person in the inpatient EMU to introduce and recruit for the study.

Inpatient epilepsy monitoring unit (EMU) address:

VUH Floor 6, Neurology/Epilepsy, 1211 Medical Center Dr, Nashville, TN 37232.

[6.0. Study Procedures] All data collection from participants' routine clinical care in this study include: Electroencephalography data from participants' inpatient admission for observational EEG monitoring at VUMC, to be collected from EPIC.

All interventions, experimental manipulations, data collection procedures, and measurements conducted for research purposes only in this study include: University of Pennsylvania Smell Identification Test™ (UPSIT®) test assessing for participant recognition of common scents on "scratch and sniff" odor cards at the beginning of the study, to be collected via REDCAP survey. Respiratory belt worn by participant as a noninvasive physical sensor applied to the surface of the body for 48 hours, to be collected via REDCAP survey. Administration of visual analog mood scales (VAMS) mood questionnaire at 24 hours and 48 hours of study timeline, to be collected via REDCAP survey. Rose scent essential oil diffusor placed in room for rose odor exposure for 24 hours between Hour 24 and 48 of study timeline.

The days and time frame of the study for participants are as follows: Day 0: In-person patient agreement to participate in study and obtainment of written informed consent. Day 1: Pre-exposure VAMS mood assessment survey, UPSIT test administration, observational EEG and respiratory belt monitoring on room air. Day 2: Observational EEG and respiratory belt monitoring with rose scent diffusor in room, post-exposure VAMS mood assessment survey.

Description of Participant Experiences:

1. When the participant agrees to take part in the study, written informed consent will be obtained by study personnel.
2. After the participant has agreed to take part in the study and informed consent has been obtained, an initial odor perception screening test using the University of Pennsylvania Smell Identification Test™ (UPSIT®) scent detection kit, a 40-item one-time test which assesses the participant's recognition of common scents like lemon, coffee, and others from a scratch and sniff pack, to measure the participant's baseline sensory intake of scents before their exposure to the rose scent. The study coordinator will instruct the participant to identify different scents from scratch and sniff cards provided by the kit. This portion of the study will be conducted in the form of a short one-on-one interview with the participant and the study coordinator, with responses recorded securely via survey in REDCAP.
3. Assessment of participants' mood during the control arm of the study will be conducted through use of a visual analogue mood scale (VAMS) collected via REDCAP. The survey will ask participants to rate their mood on various sliding scales (i.e., "happy" to "sad", "calm" to "worried") with corresponding visual representations of these emotions (i.e., "smiley face" to "frowning face").
4. Participants will then undergo their routine inpatient observational EEG monitoring for 24 hours on room air in the control arm of the study. During this time, participants will wear a respiratory belt on their upper chest for a noninvasive measure of respiratory function at baseline. Otherwise, participants will be instructed that they are free to conduct themselves as they would in any routine observational inpatient EMU stay.
5. Following the control arm, participants will undergo 24 hours of routine inpatient EEG monitoring with rose scent diffused in their room via essential oil diffusor to achieve the exposure arm of the study. Participants will continue wearing their respiratory belt on their upper chest during this branch of the study. During this time, participants will again be instructed that they are free to conduct themselves as they would in any routine observational inpatient EMU stay, the only limitation in addition to their routine clinical care being that they wear the respiratory belt superficially over their upper chest area.
6. Assessment of participants' following exposure to rose scent will be conducted through use of the visual analogue mood scale (VAMS), using the same scale and survey collection method as the pre-exposure VAMS assessment.

[7.0. Risks]

To our knowledge, there is no risk or adverse effects associated with usage of respiratory monitoring devices nor diffusers/rose odor exposure. There are small studies suggesting that rose odor exposure may have an anxiolytic effect.

[8.0. Reporting of Adverse Events or Unanticipated Problems involving Risk to Participants or Others]

All Adverse Events will be reported to the IRB as required by VHRPP policy III.L within 7 calendar days of the VU or VUMC Investigator's knowledge of the problem.

In the event of any adverse effect, Key Study Personnel will send a report to the Vanderbilt risk management team (the regulatory authority at VUMC) by logging into Vanderbilt VERITAS online portal and submitting the online report to the risk management team.

[9.0. Study Withdrawal/Discontinuation]

The main indication of withdrawal during the study would be patient themselves opting out. Other minor indication includes: diffuser or belts causing patient discomfort.

[10.0. Statistical Considerations]

The majority of patients in the EMU will be there to have medications aggressively weaned in order to capture seizure events. However, by recent historical averages, there is a roughly 2-3 patients per week at VUMC that are monitored for at least 2 days without any changes in medications. Between 60-90% of patients with known epilepsy will have epileptiform discharges on extended EEGs, therefore we can anticipate that on a 48hr EEG nearly all of the patients will have discharges to quantify. It will be less likely to observe seizures on patients without withdrawal of medications, we can estimate that 30% may have a seizure. Of these, per published reports, up to 70% of focal epilepsy patients will have associated apneas with their seizures.

Given these expectations from the extant literature, over the 16 months of enrollment, we can expect 32 patients, of which 27 will have epileptiform discharges to quantify. Of those 32 patients, 11 will have seizures where we can assess for related apneas, some patients are likely to have multiple seizures, so 15 total seizures is a conservative estimate. In addition to seizure related apneas, the record can also be analyzed for other apneas and breathing changes during the admission.

Power calculations at 80% power and alpha 5% expecting to see a 40% decrease in epileptiform discharges suggest a sample size (patient number) of 32 that we will need, which is in line with what we are expected to record over the course of this study. Our seizure related apnea analysis may be underpowered based on our expected enrollment and seizure number, if we hope to see a decrease in apnea associated with rose odor exposure of 50% then we would need 23 seizures collected.

[11.0. Privacy/Confidentiality Issues]

1. Consent will be gathered by the Key Study Personnel which includes PI Dr. William Nobis at the time of admission to the EMU. All of the above listed faculty have in depth knowledge of the research to be conducted.
2. Respiratory data will be stored, embedded with the EEG data in the same manner as all of our EEG information is stored in the EMU.
3. PHI and registration data will be stored in hospital electronic medical record (EMR) and Vanderbilt RedCap Database.

[12.0. Follow-up and Record Retention] Duration of study: 16 months. Respiratory data included with EEG and will be kept and archived per EMU protocol, with indefinite archival of information.

ELIGIBILITY:
Inclusion Criteria:

* Adult epilepsy patients over the age of 18
* Admission to the inpatient epilepsy monitoring unit (EMU) at Vanderbilt University Medical Center (VUMC)
* Undergoing observational EEG monitoring without treatment involving seizure medication changes or other interventions for at least 48 hours

Exclusion Criteria:

* Patients under the age of 18
* Patients receiving EEG monitoring without interventions from baseline for less than 48 hours
* Patients who are not receiving EEG monitoring as a part of their inpatient admission.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2026-05-08 (Estimated); Study Completion 2026-05-08 (Estimated)

PRIMARY OUTCOMES:
Number of ictal episodes | 24 hours
  Number of ictal episodes measured via EEG
Number of apneic episodes | 24 hours
  Number of brief cessations in breathing captured via respiratory belt

CONTACTS AND LOCATIONS:
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Immediately following publication. No end date.
Access Criteria: Researchers who provide a methodologically sound proposal, to achieve aims in approved proposal.

REFERENCES:
- [Background] Yilmaz Y, Turk BG, Ser MH, Sut NY, Sahin S, Yildiz EP, Bektas G, Teber ST, Tekeli H, Ozkara C. Seizure treatment with olfactory training: a preliminary trial. Neurol Sci. 2022 Dec;43(12):6901-6907. doi: 10.1007/s10072-022-06376-2. Epub 2022 Sep 6. PMID 36066675
- [Background] Valentine PA, Fremit SL, Teskey GC. Sensory stimulation reduces seizure severity but not afterdischarge duration of partial seizures kindled in the hippocampus at threshold intensities. Neurosci Lett. 2005 Nov 4;388(1):33-8. doi: 10.1016/j.neulet.2005.06.028. PMID 16039062
- [Background] Rhone AE, Kovach CK, Harmata GI, Sullivan AW, Tranel D, Ciliberto MA, Howard MA, Richerson GB, Steinschneider M, Wemmie JA, Dlouhy BJ. A human amygdala site that inhibits respiration and elicits apnea in pediatric epilepsy. JCI Insight. 2020 Mar 26;5(6):e134852. doi: 10.1172/jci.insight.134852. PMID 32163374
- [Background] O'Neal TB, Shrestha S, Singh H, Osagie I, Ben-Okafor K, Cornett EM, Kaye AD. Sudden Unexpected Death in Epilepsy. Neurol Int. 2022 Jul 18;14(3):600-613. doi: 10.3390/neurolint14030048. PMID 35893283
- [Background] Nobis W, Huffman R, Mitchell A, Hannalla M. 512 Odorant exposure decreases mortality in a Dravet Syndrome mouse model. J Clin Transl Sci. 2023;7(Suppl 1):145. Published 2023 Apr 24. doi:10.1017/cts.2023.511
- [Background] Nobis WP, Gonzalez Otarula KA, Templer JW, Gerard EE, VanHaerents S, Lane G, Zhou G, Rosenow JM, Zelano C, Schuele S. The effect of seizure spread to the amygdala on respiration and onset of ictal central apnea. J Neurosurg. 2019 Apr 5;132(5):1313-1323. doi: 10.3171/2019.1.JNS183157. Print 2020 May 1. PMID 30952127
- [Background] Nguyen MQ, Ryba NJ. A smell that causes seizure. PLoS One. 2012;7(7):e41899. doi: 10.1371/journal.pone.0041899. Epub 2012 Jul 27. PMID 22848650
- [Background] Motoki A, Akamatsu N, Fumuro T, Miyoshi A, Tanaka H, Hagiwara K, Ohara S, Kamada T, Shigeto H, Murai H. Characteristics of olfactory dysfunction in patients with temporal lobe epilepsy. Epilepsy Behav. 2021 Dec;125:108402. doi: 10.1016/j.yebeh.2021.108402. Epub 2021 Nov 12. PMID 34775249
- [Background] Lunardi MS, Lin K, Mameniskiene R, Beniczky S, Bogacz A, Braga P, Guaranha MSB, Yacubian EMT, Samaitiene R, Baykan B, Hummel T, Wolf P. Olfactory stimulation induces delayed responses in epilepsy. Epilepsy Behav. 2016 Aug;61:90-96. doi: 10.1016/j.yebeh.2016.05.022. Epub 2016 Jun 23. PMID 27344500
- [Background] Li Z, Chen L, Xu C, Chen Z, Wang Y. Non-invasive sensory neuromodulation in epilepsy: Updates and future perspectives. Neurobiol Dis. 2023 Apr;179:106049. doi: 10.1016/j.nbd.2023.106049. Epub 2023 Feb 20. PMID 36813206
- See also: Rose Scent — https://www.essentialoil.com/products/rose-oil-bulgarian?_pos=3&_sid=625f64829&_ss=r
- See also: Aroma Ace Diffuser — https://www.diffuserworld.com/store/Aroma-Acetm-MINI-Diffuser-p206368565
- See also: UPSIT Smell Test — https://sensonics.com/product/smell-identification-test/?srsltid=AfmBOopYGO_bERSXrcO_oB0rmeoqq-ueN4ZnnupMDwd9xjdatFmmQDfI